CLINICAL TRIAL: NCT05810792
Title: A Phase I/II Trial of Peri- and Postoperative Treatment With Histamine Dihydrochloride and Low-dose Interleukin-2 in Patients With Primary Resectable Pancreatic Cancer
Brief Title: Histamine Dihydrochloride and Interleukin-2 in Primary Resectable Pancreatic Cancer
Acronym: PANCEP-1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Svein Olav Bratlie, Senior surgeon, Dr Med, PhD, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANCEP-1, April 1 2020
Record Dates: First submitted 2023-03-07; First posted 2023-04-12 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Cancer; Surgery; Metastasis; Immunosuppression
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Histamine; Interleukin-2

STUDY DESIGN:
Intervention Model Description: This is a single center, open-label study in subjects with resectable pancreatic cancer. Eligible subjects will be offered treatment with histamine dihydrochloride and low-dose interleukin-2. Secondary endpoints comparing matched historical controls (DFS, OS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients receiving immunomodulating treatment (Experimental)
  Interventions: Drug: Histamine Dihydrochloride (HDC); Drug: Interleukin-2 (IL-2)

INTERVENTIONS:
Drug: Histamine Dihydrochloride (HDC) — HDC is administrated in combination with IL-2 as peri- and post-operative treatment in patients undergoing surgery. 0.5 mg HDC is administered twice daily by subcutaneous injections 1 to 3 minutes after each IL-2 injection during three 3 week cycles, with 3-week resting periods inbetween. The first treatment cycle is initated 2 weeks prior to surgery, with an additional 2-3 days rest period during the surgical procedure, before the third treatment week is initiated.
Drug: Interleukin-2 (IL-2) — IL-2 is administrated in combination with HDC during three 3 week cycles as peri- and post-operative treatment in patients undergoing surgery. IL-2 is administered twice daily as a subcutaneous injection 1 to 3 minutes prior to the administration of histamine dihydrochloride; each dose of IL-2 is 16,400 IU/kg (1µg/kg).

SUMMARY:
A key aspect of the trial is that functions of anti-neoplastic T cells and natural killer (NK) cells, may be inhibited by immunosuppressive signals from myeloid cells, in particular reactive oxygen species (ROS) produced by several subsets of myeloid cells. In cancer, such immunosuppressive cells are commonly denoted myeloid-derived suppressor cells (MDSCs), which are immature monocytes and granulocytes that impede immune-mediated clearance of malignant cells by multiple mechanisms, including the formation of immunosuppressive ROS via myeloid cell NADPH oxidase (NOX2). The presence of MDSCs within or adjacent to tumor tissue is assumed to facilitate the growth and spread of tumors and may also dampen the efficacy of cancer immunotherapies. The underlying hypothesis for this clinical trial is the administration of HDC/IL-2 will reduce surgery-induced inflammation and reduce metastasis. A phase I/II open label, single-center study of the safety, tolerability, and efficacy of peri- and postoperative therapy with histamine dihydrochloride and low-dose interleukin-2 treatment in subjects with primary pancreatic cancer.To assess the frequency and extent of adverse events associated with low dose interleukin-2 and histamine dihydrochloride when used as perioperative therapy.To determine progression free survival and overall survival following surgery, and compare with matched historical controls from the Swedish Cancer Registry.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must give written informed consent prior to initiation of therapy, in keeping with the policies of the institution.
2. Subject is a male or female age >18
3. By the surgeon´s evaluation fit for pancreatic surgery
4. Subjects must have radiologic, and or cytologic confirmation of primary pancreatic cancer

Exclusion Criteria (any of the following):

1. Class III or IV cardiac disease, hypotension or severe hypertension, vasomotor instability, serious or uncontrolled cardiac dysrhythmias (including ventricular arrhythmias) at any time, acute myocardial infarction within the past 6 months, active uncontrolled angina pectoris or symptomatic arteriosclerotic peripheral blood vessel disease.
2. History of uncontrolled seizures, severe central nervous system disorders, or psychiatric disability thought to be clinically significant in the opinion of the Investigator and adversely affecting compliance to protocol.
3. Any other condition or symptoms preventing the patient from entering the study, according to the PI's judgement.
4. A woman of childbearing potential (WOCBP) must agree to comply with using an effective contraceptive method for the duration of the treatment (a WOCBP is a sexually mature woman who is not surgically sterile or has not been naturally postmenopausal for at least 12 consecutive months). Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly. Local laws and regulations may require use of alternative and/or additional contraception methods. One of the highly effective methods of contraception listed below is required during study duration and until the end of relevant systemic exposure, defined as 5 months after the end of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Treatment-Emergent Adverse Events as assessed by NCI-CTCAE | When the first 14 patients have undergone one full 3-week cycle with HDC/IL-2 (approximately 18 months after trial start)
  Incidence and severity grade of adverse events occuring during and after treatment will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0.

SECONDARY OUTCOMES:
Overall survival | 24 months
  Comparing matched historical controls from national registry
Disease free survival | 24 months
  Comparing matched historical controls from national registry
Changes in Natural killer cell subsets in blood | Change from pre-surgical levels to levels during the post-surgical week
  Changes in NK cell number and expression of activation markers during surgery
Changes in T cell subsets in blood | Change from pre-surgical levels to levels during the post-surgical week
  Changes in T cell number and expression of activation markers during surgery
Changes in Myeloid cell populations | Change from pre-surgical levels to levels during the post-surgical week
  Changes in myeloid cell number and markers of activation and inhibition
Tumor infiltrating lymphocytes and tumor infiltrating myeloid cells | immediately after the surgery
  Tumor pieces removed during surgery will be assessed for immune populations
Carbohydrate antigen 19-9 | 12 months
  Serum CA 19-9 levels are monitored as a biomarker for disease recurrance

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Muth, Study Director — Västra Götalandsregionen, Sahlgrenska University Hospital

IPD SHARING:
Plan to Share IPD: No